CLINICAL TRIAL: NCT04484155
Title: Minimally Invasive Micro Sclerostomy: First in Man (FIM) Safety and Preliminary Performance Study
Brief Title: Minimally Invasive Micro Sclerostomy: Safety and Preliminary Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMS-072-51
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally invasive micro sclerostomy (MIMS) (Experimental): create a drainage channel at the sclera-corneal junction
  Interventions: Device: Minimally Invasive Micro Sclerostomy (MIMS)

INTERVENTIONS:
Device: Minimally Invasive Micro Sclerostomy (MIMS) — The System is a surgical device, designed to create a drainage channel at the sclera-corneal junction . The drainage channel is created by a Stainless Steel surgical tool.

SUMMARY:
Eligible Glaucoma patients will undergo pre-surgery examination including:

medicines list, blood tests and ECG. On surgery day: intraocular pressure (IOP) will be measured. Then a sub-conjunctival injection of Mitomycin C will be administered .

The Minimally Invasive Micro Sclerostomy (MIMS) procedure is designed to create a drainage channel at the sclera-corneal junction by penetrating through the wall [scleral tissue] . MIMS procedure may be combined with cataract surgery.

Patients will be followed up to 24 weeks post operation.

DETAILED DESCRIPTION:
Eligible patients will have ECG and blood test up to 30 days prior to the MIMS procedure.

Description of MIMS procedure:

on surgery day, intraocular pressure (IOP) will be measured. Then a sub-conjunctival injection of Mitomycin C will be administered .

creating drainage channel at the sclera-corneal junction by penetrating through the wall [scleral tissue].MIMS procedure may be combined with cataract surgery.

Post-operatively the patient will be treated with dexamethasone-neomycin drops for at least one month.

Patients will be followed up to 24 weeks post operation.

The following measurements will be included:

* Intra Ocular Pressure (IOP)
* Best Corrected Visual Acuity (BCVA)
* Slit Lamp Biomicroscopic evaluation
* Anterior Segment Optical coherence tomography (OCT)
* Fundus Examination

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* End stage Primary open-angle glaucoma,pseudoexfoliation glaucoma or pigmentary glaucoma in the study eye
* Optic nerve appearance characteristic of glaucoma in the study eye
* Best-corrected visual acuity (BCVA) with ETDRS charts ≤ 6/60
* Patient is treated with 0 to 5 hypotensive medications in the study eye
* Unsatisfactory IOP (≥ 21 mmHg) at the screening visit in the study eye
* If cataract is not present - Shaffer grade ≥ III in all four angle quadrants in the study eye
* Subject is able and willing to attend all scheduled follow-up exams
* Subject understands and signs the informed consent

Exclusion Criteria:

* Ocular conditions with a poorer prognosis in the fellow eye than in the study eye
* Closed angle forms of glaucoma in either eye unless scheduled for cataract surgery immediately prior to the MIMS procedure or the study eye is pseudophakic with PCIOL.
* Congenital or developmental glaucoma in either eye
* Other secondary glaucoma (such as neovascular, uveitic, lens-induced, trauma-induced, or glaucoma associated with increased episcleral venous pressure) in the study eye
* Peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities in the study eye
* Subject has history of penetrating keratoplasty (PKP)
* Any previous surgery in the study eye (except for clear corneal cataract surgery) where the conjunctiva is not intact and elastic.
* Any ocular disease or history in study eye such as severe dry eye, active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, and ocular pathology that may interfere with accurate IOP measurements
* Prior surgery for an ab-interno or ab-externo device implanted in or through the Schlemm's canal in the study eye.
* Use of oral hypotensive medication for glaucoma for treatment of the fellow eye
* Best-corrected visual acuity worse than 20/50 (Snellen equivalent) in the fellow eye
* History of idiopathic or autoimmune uveitis in either eye
* Severe trauma in study eye
* active iris neovascularization, previous cyclodestructive procedure, prior scleral buckling procedure, presence of silicone oil
* Vitreous present in anterior chamber, prior vitrectomy or virteous hemorrhage in study eye
* Aphakia
* Prior vitreoretinal surgery in study eye
* Clinically significant ocular inflammation or infection within 90 days prior to screening
* Unable to discontinue use of blood thinners in accordance with surgeon's standard preoperative instructions
* Uncontrolled systemic disease that in the opinion of the investigator would put the subject's health at risk and/or prevent the subject from completing all study visits
* Current participation or participation in another investigational drug or device clinical trial within the last 30 days before screening visit
* Pregnant or lactating women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Event | 12 weeks
  Overall incidence of serious adverse events
Drainage Channel Creation | Index procedure day
  Ability to successfully perform a drainage channel

SECONDARY OUTCOMES:
Serious Adverse Event | 24 Weeks
  Overall incidence of serious adverse events
Intraocular Pressure | 24 Weeks
  Intraocular Pressure between 6 mmHg and 20 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Agarwal Eye Hospital Ltd., Chennai, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geffen N, Kumar DA, Barayev E, Gershoni A, Rotenberg M, Zahavi A, Glovinsky Y, Agarwal A. Minimally Invasive Micro Sclerostomy (MIMS) Procedure: A Novel Glaucoma Filtration Procedure. J Glaucoma. 2022 Mar 1;31(3):191-200. doi: 10.1097/IJG.0000000000001955. PMID 34731867